CLINICAL TRIAL: NCT02488291
Title: Effect of 0.5µg/ml Sufentanil and Ropivacaine Towards Pregnant Women and Fetus in Analgesia Labor
Brief Title: Effect of Sufentanil and Ropivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zeyong Yang, Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPMCH
Record Dates: First submitted 2015-06-20; First posted 2015-07-02 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia Complications
Keywords: Epidural; Analgesia labor; Perinatal; anesthesia
MeSH Terms: interventions — Sufentanil; Ropivacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5 sufentanil (Experimental): 0.5µg/ml sufentanil, 0.1% ropivacaine for 6ml/h
  Interventions: Drug: 0.5µg/ml sufentanil; Drug: 0.1% ropivacaine
- 0.25 sufentanil (Experimental): 0.25µg/ml sufentanil, 0.1% ropivacaine for 6ml/h
  Interventions: Drug: 0.25 sufentanil; Drug: 0.1% ropivacaine

INTERVENTIONS:
Drug: 0.25 sufentanil — with different dosage
  Other Names: opiods
  Arms: 0.25 sufentanil
Drug: 0.5µg/ml sufentanil — 0.5µg/ml sufentanil
  Other Names: opiods
  Arms: 0.5 sufentanil
Drug: 0.1% ropivacaine — 0.1% ropivacaine
  Other Names: Local Anesthetics

SUMMARY:
The investigators study the efficacy of epidural sufentanil/ropivacaine for analgesia labor in primiparas so as to decrease perinatal complications of analgesia labor.

DETAILED DESCRIPTION:
A prospective study of 120 full-term parturients receiving labor analgesia were randomly assigned into 2 groups: the 0.5Sufen group (N=60), the 0.25Sufen group (N=60).

ELIGIBILITY:
Inclusion Criteria:

1. Patients had regular prenatal examinations at the outpatient clinic;
2. They were between 25 to 35 years of age)
3. They had a gestational age ≥37 weeks and < 42 weeks;
4. They had an estimated fetal weight ≥ 2,500 g and < 4,200 g.

Exclusion Criteria:

* a history of spinal surgery,
* platelet count <100×109 /L ,
* coagulation disorder,
* sensorimotor disorder of lower extremity,
* leg pain,
* puncture point infection,
* heart disease history,
* pulmonary disease,
* liver and renal function disorder and
* a history of neuropsychiatry drugs.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
VAS(visual analog pain score) | 1 year
  comparison with two groups

CONTACTS AND LOCATIONS:
Overall Officials: Zeyong Yang, M.D., Principal Investigator — Fudan University, Shanghai Jiaotong University

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02488291/SAP_000.pdf